CLINICAL TRIAL: NCT04735198
Title: Effectiveness of Prophylactic Cholecystectomy in Patients With Midgut Neuroendocrine Tumor (Jejunum, Ileum or Proximal Colon) Who Require Primary Tumor Surgery. Randomized, Proof of Concept Clinical Trial.
Brief Title: Prophylactic Cholecystectomy in Midgut NETs Patients Who Require Primary Tumor Surgery.
Acronym: TNE-IDC-COLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Ricardo Frago Montanuy, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR348/20
Record Dates: First submitted 2021-01-21; First posted 2021-02-03 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Midgut Carcinoid Tumor; Biliary Stones
Keywords: Neuroendocrine tumor; prophylactic cholecystectomy; Biliary stone disease
MeSH Terms: conditions — Cholecystolithiasis; Neuroendocrine Tumors | interventions — Colectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Active Comparator): Patients with midgut neuroendocrine tumor who will undergo only primary tumor surgery.
  Interventions: Procedure: Primary tumor surgery
- Control group (Experimental): Patients with midgut neuroendocrine tumor that will undergo through primary tumor surgery combined with prophylactic cholecystectomy.
  Interventions: Procedure: Primary tumor surgery; Procedure: Primary tumor surgery (bowel resection) combined with prophylactic cholecystectomy

INTERVENTIONS:
Procedure: Primary tumor surgery — Large bowel resection.
  Other Names: Bowel resection
Procedure: Primary tumor surgery (bowel resection) combined with prophylactic cholecystectomy — Large bowel resection combined and cholecystectomy.
  Other Names: prophylactic cholecystectomy.
  Arms: Control group

SUMMARY:
The investigators want to study the effectiveness of prophylactic cholecystectomy in patients with midgut neuroendocrine tumor (jejunum, ileum or proximal colon) who require primary tumor surgery. When patients are diagnosed and are tributary to surgical treatment, the tumor might compromise vascularization, and patients need an extensive bowel resection. The patients might also receive medical treatment with somatostatin analogs. The combination of extensive bowel resection and medical treatment might increase gallbladder stones, but patients might not develop biliary stone disease, as in the general population, where 20% of the population have gallbladder stones but only a 10 to 15 % of the population will develop symptoms.

The idea comes from the lack of literature about the incidence of biliary Stone disease in patients with midgut NET tumors.

It's a multicentric, open-label and randomized clinical trial to evaluate the incidence of biliary stone disease in patients with midgut NET who require primary tumor surgery combined or not to cholecystectomy.

Our hypothesis suggests that patients with midgut neuroendocrine tumor who require primary tumor resection without the combination of prophylactic cholecystectomy do not have an increased incidence of biliary stone disease two years after the surgery, regardless of treatment with SSA.

DETAILED DESCRIPTION:
Title: Effectiveness of prophylactic cholecystectomy in patients with midgut neuroendocrine tumor (jejunum, ileum or proximal colon) who require primary tumor surgery. Randomized, proof of concept clinical trial.

Background: The prevalence of midgut NET has increased due to advances in diagnostic tests and its indolent course. When patients are diagnosed, they might be tributary to surgical treatment requiring an extensive bowel resection, and medical treatment with somatostatin analogs. Both treatments are related with gallbladder stone formation. The ENETS and NANETs recommend prophylactic cholecystectomy in patients with midgut NET who require primary tumor surgery, However, there is a lack of scientific evidence reinforcing this recommendation.

Objectives: The main objective is to evaluate the cumulated incidence rate of biliary stone disease in patients with midgut NET who require primary tumor resection, two years after the surgery.

Design: It's a multicentric, open-label and randomized clinical trial. Patients will be recruited from the General Surgery Services of the six Hospitals participating in the study. Patients must fullfill inclusion and exclusion criteria.

It is expected to recruit a maximum of one hundred patients in two years (50 per group). Patients will be randomly assigned into the Experimental group (primary tumor resections) or Control group (primary tumor resections combined with cholecystectomy). The investigators will follow up patients until week 104 after surgery (8 visits).

ELIGIBILITY:
Inclusion Criteria:

* Patients must grant the informed consent written, signed and dated.
* Male or female older than 18 years old.
* Radiological or histological diagnose of midgut NET that can be treated with surgery.
* In case of female with childbearing age (time between menarche and menopause), a pregnancy test with negative result.
* Neuroendocrine tumors located in any of the aforementioned locations.
* Presence or not of distant metastasis.
* Presencié or not of gallstones.
* Capacity of follow up.

Exclusion Criteria:

* Neuroendocrine tumors which are not located in jejunum or ileum (bronchial, gastric, pancreatic, descending colon, sigma or rectum.).
* Patients that have gone through a previous bowel resection.
* Patients with previous cholecystectomy.
* Pacients with biliary stone disease.
* Patients who are candidate to liver resection or liver transplant.
* Patients with a gallbladder polyp bigger than 6 mm.
* Pacients with one gallbladder sessile polyp, presence of more than one polyp or patients older than 50 years old with a polyp.
* Refusal to participate.
* Patients with previous history of malignant neoplasms in the last 5 years, except skin basal cell carcinoma, "in situ" cervical carcinoma or in situ carcinoma found in a polyp removed with a colonoscopy.
* Medical criteria that doesn't consider the patient a candidate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the rate of biliary stone disease associated to patients with midgut NET that have gone through primary tumor surgery. | Two years after the surgery
  Incidence of biliary stone disease in patients with midgut NET who requiere primary tumor surgery

SECONDARY OUTCOMES:
To assess the incidence of post-operative complications until day 28 +/- 3 (1 Month) after the surgery. | One month after the surgery
  Postoperative complications according Clavien-Dindo classification
To assess the incidence of: anastomotic dehiscence, wound infection, reoperation. | One month after the surgery
  Specific complications
To evaluate the incidence of gallstone in patients who require a bowel resection and/or ileocecal junction resection. | Two years after the surgery
  choledochal lithiasis or cholelithiasis
To evaluate de incidence of gallstones in patients who will receive medical treatment with SSA | Two years after the surgery
  choledochal lithiasis or cholelithiasis according medical treatment
To describe bowel movements of patients after the surgery. | Two years after the surgery
  Gastrointestinal Quality of Life Index (GIQLY);Minimum value of 0 (the worst health state) and a maximum of 100 (best health state)
To compare quality of life in patients who went through a prophylactic cholecystectomy against those who did not. | Two years after the surgery
  Health related Quality of life 15 D (HRQoL 15D);There are 15 areas with a minimum value of 0 (the worst health state) and a maximum of 100 (best health state) 15D

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Frago Montanuy, Principal Investigator — Hospital Universitari de Bellvitge
Locations (6):
- Spain (6):
  - Hospital Universitari Trias i Pujol, Badalona, Barcelona
  - IDIBELL, Hospital Universitari de Bellvitge., Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Instituto Catalán de Oncología, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
That's not decided yet